CLINICAL TRIAL: NCT02340403
Title: Exploration by NMR Spectroscopy of the Choline Concentrations in the Insular Cortex of Patients Suffering of Neuropathic Pain Induced by Oxaliplatin
Acronym: INSULOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-0217; 2013-A01588-37 (Registry Identifier: 2013-A01588-37)
Record Dates: First submitted 2015-01-08; First posted 2015-01-16 (Estimated); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Neuropathy; Painful
Keywords: Neuropathy; Oxaliplatin; Insula; choline
MeSH Terms: conditions — Pain | interventions — Magnetic Resonance Spectroscopy

ARMS (2):
- Oxaliplatin and neuropathic pain (Experimental): The objective of this study is to demonstrate a significant increase in choline concentration in the insular cortex of patients with an oxaliplatin induced neuropathy. Other objectives will assess the correlation between metabolite concentrations in the insular cortex and frequency / intensity of pain and neuropathic symptoms, cold and heat-induced pain and comorbidities (anxiety, pain, quality of life).
  Interventions: Procedure: NMR Spectroscopy
- Oxaliplatin without neuropathic pain (Other): The objective of this study is to demonstrate a significant increase in choline concentration in the insular cortex of patients with an oxaliplatin induced neuropathy. Other objectives will assess the correlation between metabolite concentrations in the insular cortex and frequency / intensity of pain and neuropathic symptoms, cold and heat-induced pain and comorbidities (anxiety, pain, quality of life).
  Interventions: Procedure: NMR Spectroscopy

INTERVENTIONS:
Procedure: NMR Spectroscopy

SUMMARY:
Neurotoxic chemotherapy, including oxaliplatin, are responsible for very disabling neuropathic pain that can last for months or even years after the end of chemotherapy. Currently, there is no effective neuroprotective treatment to prevent or relieve this pain. The only strategy is the reduction of oxaliplatin doses or premature discontinuation of therapy, with the risk of burdening the prognosis for remission. Thus, a better understanding of the pathophysiology of these iatrogenic neuropathies appears necessary in order to discover new potential therapeutic targets.

Preclinical works were able to demonstrate important metabolic changes in certain brain structures in an animal model of oxaliplatin-induced neuropathy. A significant increase of choline concentration has been found in the posterior insular cortex of neuropathic animals compared with control animals. Furthermore, the concentrations of choline were positively correlated to nociceptive thresholds. Thus, neuropathic pain induced by oxaliplatin would involve the posterior insular cortex and would be associated with an increase in choline concentration at this level. Clinical translation of these preclinical results is feasible in practice since choline concentration can be determined in the brain by non-invasive magnetic resonance spectroscopy.

DETAILED DESCRIPTION:
The objective of this study is to demonstrate a significant increase in choline concentration in the insular cortex of patients with an oxaliplatin induced neuropathy. Other objectives will assess the correlation between metabolite concentrations in the insular cortex and frequency / intensity of pain and neuropathic symptoms, cold and heat-induced pain and comorbidities (anxiety, pain, quality of life).

ELIGIBILITY:
Inclusion Criteria:

* Oxaliplatin treated patient and suffering from neuropathic pain

  * Chemotherapy (oxaliplatin based) ended
  * Pain VAS ≥ 3/10, 1 month after the chemotherapy end
  * DN4 interview score ≥ 3/7, 1 month after the chemotherapy end
* Oxaliplatin treated patient without neuropathic pain

  * Chemotherapy (oxaliplatin based) ended
  * Pain VAS < 3/10, 1 month after the chemotherapy end
  * DN4 interview score < 3/7, 1 month after the chemotherapy end
* All patients

  * right-handed
  * No contrindication to MRI
  * Free, written and informed consent
  * Affiliated to the french health system
  * Effective contraception for male or female of childbearing age
  * Performance score (WHO) ≤ 2

Exclusion Criteria:

* Age < 18
* Left-handed
* BMI > 30 kg/m²
* Amputees of all or part of an upper limb
* Diabetic patient
* Painful events scheduled after enrollment (eg. surgical resection)
* Neurological diseases (eg Parkinson's disease, stroke, migraine, fibromyalgia ...)
* Chronic pain history before chemotherapy
* Analgesic treatment being other than paracetamol and weak opioids
* Alcohol consumption >3 units/day (30 g/day) for men and >2 units/day (20 g/day) for women
* Any unbalanced progressive disease (hepatic failure, renal impairment (creatinine clearance <30 mL/min), respiratory failure, congestive heart failure, myocardial infarction within the past 6 months ...)
* All active cancer
* Patient with a pacemaker, a cochlear implant, metal implants, or any other magnetic element
* Claustrophobia
* Pregnant or lactation
* Legal incapacity (person deprived of liberty or guardianship)
* Psychological, social, family or geographical reasons incompatible with the study
* Already included in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-03-09 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
Choline concentration assessed by NMR spectroscopy in the posterior insula | 1 month after chemotherapy end

SECONDARY OUTCOMES:
Metabolite concentrations assessed by NMR spectroscopy in the posterior insula | 1 month and 6 months after chemotherapy end
  Metabolite (choline, myo-inositol, N-acétylaspartate, créatine, glutamate/glutamine, lactate and taurine)
Pain intensity (VAS and BPI questionnaire) | 1 month and 6 months after chemotherapy end
  (VAS and BPI questionnaire)
Neuropathic pain diagnostic 9DN4 interview questionnaire) | 1 month and 6 months after chemotherapy end
Neuropathic pain intensity (NPSI questionnaire) | 1 month and 6 months after chemotherapy end
  NPSI questionnaire
BPI questionnaire | 1 month and 6 months after chemotherapy end
Quantitative sensory threshold (cold, heat, vibration) | 1 month and 6 months after chemotherapy end
Neuropathy grade | 1 month and 6 months after chemotherapy end
Anxiety and depression symptoms (HADS questionnaire) | 1 month and 6 months after chemotherapy end
  HADS questionnaire
Intensity of chemotherapy-induced peripheral neuropathy (CIPN20 questionnaire) | 1 month and 6 months after chemotherapy end
  CIPN20 questionnaire
Health related quality of life (QLQ-C30 questionnaire) | at 1 month and 6 months after chemotherapy end
  (QLQ-C30 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France